CLINICAL TRIAL: NCT02358291
Title: Microendoscopic Discectomy Vs Transforaminal Endoscopic Lumbar Discectomy Vs Open Discectomy for the Treatment of Lumbar Disc Herniation
Brief Title: Microendoscopic Discectomy Vs Transforaminal Endoscopic Lumbar Discectomy Vs Open Discectomy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Kun Wang, Kun Wang, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WANG-8808-KUN
Record Dates: First submitted 2015-01-26; First posted 2015-02-06 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- open discectomy (Active Comparator): patients diagnosed as lumbar disc herniation undergoing open simple discectomy(OD)
  Interventions: Procedure: microendoscopic discectomy; Procedure: transforaminal endoscopic lumbar discectomy
- microendoscopic discectomy (Active Comparator): patients diagnosed as lumbar disc herniation undergoing microendoscopic discectomy(MED)
  Interventions: Procedure: open discectomy; Procedure: transforaminal endoscopic lumbar discectomy
- transforaminal endoscopic discectomy (Active Comparator): patients diagnosed as lumbar disc herniation undergoing transforaminal endoscopic lumbar discectomy(TELD)
  Interventions: Procedure: open discectomy; Procedure: microendoscopic discectomy

INTERVENTIONS:
Procedure: open discectomy — The open discectomy, will be performed under general anesthesia in the prone position with horizontal. The level of the spine indicated for surgical treatment will be identified with the aid of fluoroscopy. An incision is made about the dorsal disc level involved with dissection of the paravertebral muscles on the side of disc herniation. After laminectomy and resection of part of the yellow ligament, partial discectomy is done under direct vision.
  Arms: microendoscopic discectomy; transforaminal endoscopic discectomy
Procedure: microendoscopic discectomy — Microendoscopic discectomy combines standard lumbar microsurgical techniques with endoscope, enabling surgeons to successfully address free-fragment disc pathologic factors and lateral recess stenosis.
  Arms: open discectomy; transforaminal endoscopic discectomy
Procedure: transforaminal endoscopic lumbar discectomy — transforaminal endoscopic lumbar discectomy removes the intervertebral disc portion through the intervertebral foramen
  Arms: microendoscopic discectomy; open discectomy

SUMMARY:
In our study, a multicenter randomized controlled，single blind trial will be performed to evaluate the effectiveness and safety of these three procedures for the treatment of symptomatic lumbar disc herniation.

DETAILED DESCRIPTION:
Lumbar disc herniation (LDH) is one of the most common diseases in the department of orthopedics, which produced medical and economic burdens to families and society. In spite, the majority of the patients with disc herniation can be relieved or even cured via conservative treatment; there are still a considerable number of invalid patients who eventually still need to be undergoing a surgical operation treatment. Three main methods for intervertebral disc surgery are adopted in our routine work. One procedure is Open Discectomy (OD), which has been always a gold standard for treatment of LDH. And the other two procedures are Microendoscopic Discectomy (MED) and Transforaminal Endoscopic Lumbar Discectomy (TELD) respectively. MED and TELD have been developed as alternatives to OD. OD can compress the nerve root or spinal cord through removal of the protrusion. However, it destroys the rear structure of spine, causing segmental instability and long-term distress. Compared with OD, MED and TELD procedures are smaller incisions or less dissection (or both), lower blood loss, less postoperative pain, shorter hospitalisation and earlier return to work. However, the steep learning curves of MID inhibit the development of surgery specialists; for example, optimal surgical management requires many years of experience. These deficiencies need more educational effort at a higher priority than accorded so far. There are inconsistent outcomes about the efficacy and safety in the previous studies; all of the recent researches do not yield conclusive results.

ELIGIBILITY:
Inclusion Criteria:

1. All forms of disc herniation were included in the study
2. History of concordant radicular leg pain refractory to conservative treatment for longer than 6 months
3. Leg pain must be greater than back pain

Exclusion Criteria:

1. cauda equine syndrome,
2. progressive neurologic deficit,
3. bilateral lower extremity symptoms,
4. low back pain more than leg pain
5. Systemic infection or localized infection at the anticipated entry needle site
6. combined with lumbar infection, fracture of lumbar vertebra, tumor, Ⅱ°and above spondylolisthesis, lumbar spinal stenosis, lumbar scoliosis is larger than 15 degree
7. with severe heart, brain, lungs, and other organs disease or mental illness
8. History of opioid abuse or patients currently on long acting opioid
9. History of the operation on lumbar
10. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index(ODI) | up to 104 weeks
  Oswestry Disability Index (ODI) -> The Oswestry Disability Index (ODI) is one of the principal condition-specific outcome measures used in the management of spinal disorders. The ODI is the most commonly outcome measures in patients with low back pain. Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. If the FIRST statement is marked, the section score = 0, If the LAST statement is marked, it = 5. 0 is the best outcome and 50 is the worst The ODI is the most commonly outcome measures in patients with low back pain. Each of the 10 items is scored from 0 - 5. The maximum score is therefore 50. If the FIRST statement is marked, the section score = 0, If the LAST statement is marked, it = 5. 0 is the best outcome and 50 is the worst outcome

SECONDARY OUTCOMES:
visual analogue scale(VAS) | up to 104 weeks
  Pain Score - Visual Analog Scale (VAS) -> minimum value=0 and maximum value=10, higher values represent a worse outcome and zero is a better outcome
The generic health survey on the Short Form-36(SF-36) | up to 104 weeks
  The scale was used to evaluate the quality of life
Complications survey | up to 104 weeks
  Complications of surgery including mortality and common: thrombosis; surgical site and other infections; recurrent disc herniation; dural tear; nerve root injury

CONTACTS AND LOCATIONS:
Overall Officials: Wu Xiaotao, MD, Study Director — Zhangda hospital,Southeast university

REFERENCES:
- [Result] Liu WG, Wu XT, Guo JH, Zhuang SY, Teng GJ. Long-term outcomes of patients with lumbar disc herniation treated with percutaneous discectomy: comparative study with microendoscopic discectomy. Cardiovasc Intervent Radiol. 2010 Aug;33(4):780-6. doi: 10.1007/s00270-009-9720-6. Epub 2009 Oct 15. PMID 19830485
- [Result] Wu X, Zhuang S, Mao Z, Chen H. Microendoscopic discectomy for lumbar disc herniation: surgical technique and outcome in 873 consecutive cases. Spine (Phila Pa 1976). 2006 Nov 1;31(23):2689-94. doi: 10.1097/01.brs.0000244615.43199.07. PMID 17077737